CLINICAL TRIAL: NCT05418686
Title: Study Of Colchicine Resistance In Familial Mediterranean Fever
Acronym: COLCHI-RESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP211442
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Mediterranean Fever; Colchicine Resistance
Keywords: Familial mediterranean fever; Colchicin-resistant; Drug compliance; Microbiota; Drug resistance; clostrioides difficile; interleukin-1; second-line therapy.
MeSH Terms: conditions — Brucellosis; Familial Mediterranean Fever; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colchicine-resistant Familial Mediterranean Fever patients (Experimental)
  Interventions: Biological: Capillary colchicine dosage in colchicine-resistant Familial Mediterranean Fever patients.

INTERVENTIONS:
Biological: Capillary colchicine dosage in colchicine-resistant Familial Mediterranean Fever patients. — * Adherence to colchicine therapy will be assessed by the Girerd questionnaire (6 questions ) completed by the patient at the inclusion visit.
  * A blood sample (8ml) is taken, including a haemogram, CRP and creatinine and proteinuria.
  * Standard on-site stool analysis for C. difficile toxin.
  For research purposes, samples of:
  * Stool. If the patient is unable to produce stools on the day of the visit, a collection kit with 2 tubes containing a preservative will be given to him/her as well as a stamped envelope to take the sample at home and send it by post within 10 days according to a validated procedure.
  * A strand of hair with the diameter of a pencil and a minimum length of 2 cm, in the region of the posterior vertex.
  * In patients with baldness or bleached hair only: pubic and/or axillary hair, a pencil-sized strand.
  * Additional blood (5ml) and urine (2ml) samples for colchicine determination.

SUMMARY:
Five to 10% of familial mediterranean patients are considered colchicine-resistant (i.e. patients with a persistent inflammatory syndrome, despite taking the maximum tolerated dose of colchicine daily). The recommended treatment in this case is a subcutaneous anti-interleukin 1 biotherapy (anakinra or canakinumab). These treatments are expensive (1,000 to 12,000 euros/month).

However, for a patient to be considered colchicine-resistant, compliance with the treatment must be verified. Furthermore specific activation of the pyrin inflammasome by Clostrioides difficile toxin and the overrepresentation of these bacteria in the stools of our patients led us to systematically search for them in our resistant patients. The demonstration of the involvement of C. difficile in the imbalance of the disease has not yet been published.

The colchiresist study aim to better characterize colchicine-resistance by confirming good compliance to treatment with colchicine hair measurement and by looking for clostrioides infection or intestinal dysbiosis.

DETAILED DESCRIPTION:
Patients meeting the criteria for colchicine resistance will be included in a follow-up visit.

* Adherence to colchicine therapy will be assessed by the Girerd questionnaire completed by the patient at the inclusion visit.
* A blood test is performed including a haemogram, CRP and SAA, creatinine and proteinuria.
* a standard stool analysis on site to look for C. difficile toxin.

For research purposes, samples of:

* Stool.
* A strand of hair with the diameter of a pencil and a minimum length of 2 cm, in the region of the posterior vertex, where the growth and integration are relatively constant to avoid variability.
* In patients with baldness or bleached hair only: pubic and/or axillary hair will be taken, The samples will then be processed without segmentation.
* Additional blood (5ml) and urine (2ml) samples for colchicine dosage. The patient's participation ends after this visit

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Age ≥ 12 years with no upper age limit -Patients with familial Mediterranean fever (FMF) meeting international criteria for the disease (Livneh criteria) and carrying 2 pathogenic mutations in the MEFV gene.

Patients considered colchicine-resistant according to EULAR criteria reviewed by an expert consensus:

* Persistence of signs of activity (at least one attack per month for at least 3 months) despite taking the maximum tolerated dosage of colchicine.
* Persistence of a biological inflammatory syndrome after exclusion of other causes and despite taking a maximum tolerated dosage of colchicine.
* Signature of an informed consent by the patient (or his parents if under 18 years of age)
* Patients affiliated to a social security system

Exclusion Criteria:

- Patients participating in another interventional trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Amount of colchicine measured in the first 2 cm of hair from the scalp of an FMF patient considered colchicine resistant or from pubic hair in patients with bald or colored hair, which corresponds to the average compliance of the last 2 months of intake | Through study completion, an average of 18 months
  To assess 2-month compliance with colchicine in patients with FMF considered resistant via capillary drug dosage

SECONDARY OUTCOMES:
Correlation between the amount of colchicine measured in the hair and the blood and urine levels of colchicine attesting to the last days' intake. | Through study completion, an average of 18 months
  To study blood and urine colchicine dosage in FMF patients considered resistant to colchicine
Correlation between capillary colchicine dosage and colchicine compliance assessed with the 6-item GIRERD | Through study completion, an average of 18 months
  Compare hair dosing to self-reported compliance
Composition of the fecal microbiota (search for an overrepresentation of clostridiae) in colchicine-resistant patients patients with colchicine resistance | Through study completion, an average of 18 months
  Studying the composition of the fecal microbiota in colchicine-resistant FMF patients
Testing for clostridioides difficile toxin B in colchicin-resistant patients | Through study completion, an average of 18 months
  Testing colchicine-resistant FMF patients for clostridioides difficile toxin to rule out chronic asymptomatic carriage
Dosage of proinflammatory cytokines IL1, IL6, IL18, TNFa and il1Ra. | Through study completion, an average of 18 months
  Study blood levels of proinflammatory cytokines in colchicine-resistant patients, in particular IL1 and il1RA
Percentage of patients for whom a prescription of anti-IL-1 biotherapy could have been avoided (i.e. poor compliance with Colchicine and/or Clostrioides Difficile infection) | Through study completion, an average of 18 months
  Determine the percentage of patients labeled colchicine resistant who were actually noncompliant or chronically infected with pyrin-activating bacteria like clostridioides difficile

CONTACTS AND LOCATIONS:
Overall Officials: Léa SAVEY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine Interne. Hôpital Tenon, 4 Rue de la Chine, Paris, France

IPD SHARING:
Plan to Share IPD: No